CLINICAL TRIAL: NCT05171296
Title: Noninvasive Hemoglobin Monitoring by Spectrophotometry (SpHb) in Blunt Abdominal Trauma Patients for Conservative Management
Brief Title: Noninvasive Hemoglobin Monitoring by Spectrophotometry in Blunt Abdominal Trauma Patients for Conservative Management
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FMASU R 177 / 2021
Record Dates: First submitted 2021-12-10; First posted 2021-12-28 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Intensive Care Unit
Keywords: massimo

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — complete blood count
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- abdominal trauma patients: blunt abdominal trauma patients planned for conservation.

SUMMARY:
We aimed to study the efficacy of Noninvasive Hemoglobin Monitoring by Spectrophotometry in monitoring hemoglobin level in trauma patients for conservative management.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I to III, of either sex, 18 -80 years of age, non-sedated non-intubated patients who will be admitted to Ain Shams university hospital - surgical intensive care unit, after blunt abdominal trauma planned for conservation.

Exclusion Criteria:

* Patients with fever, hypothermia, history of a neurological, psychiatric, dementia or, who are taking psychotropic drugs Patients with unstable hemodynamic status, and unconscious patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who will be admitted to Ain Shams university hospital - surgical intensive care unit, after blunt abdominal trauma planned for conservation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-08-22 (Estimated); Study Completion 2022-08-22 (Estimated)

PRIMARY OUTCOMES:
accuracy of hemoglobin measured by the noninvasive device. | 3 months
  accuracy of hemoglobin measured by the noninvasive hemoglobin test device (Radical-7®; Masimo Corp., Irvine, CA) in comparison with standard CBC that is assayed on Coulter LH 750 Cell Counter (Beckman Coulter Corporation, Florida, USA), using reagents supplied by the company in patients suffering frm blunt abdominal trauma aditted to ICU for observation.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt